CLINICAL TRIAL: NCT03542929
Title: Acute Whole Body Vibration Decrease the Glucose Levels in Elderly Diabetic Women
Brief Title: Acute Whole Body Vibration Change the Glycemic and Lactate Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maíra F Pessoa (Other)
Responsible Party: Sponsor-Investigator, Maíra F Pessoa, Clinical Professor, Universidade Federal de Pernambuco
Organization: Universidade Federal de Pernambuco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Whole body vibration glucose
Record Dates: First submitted 2018-04-12; First posted 2018-05-31 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A researcher was performed the interventional protocol and a different researcher was made the evaluations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy elderly (Active Comparator): healthy elderly were use the Whole body vibration intervention during 10 minutes
  Interventions: Device: whole body vibration
- diabetic elderly (Experimental): diabetic elderly were use the Whole body vibration intervention during 10 minutes
  Interventions: Device: whole body vibration

INTERVENTIONS:
Device: whole body vibration — whole body vibration training on a vibrating platform with healthy elderly and diabetic elderly

SUMMARY:
The type II diabetes is characterized by high levels of blood glucose followed by excessive insulin release so that the target cells become less sensitive and develop insulin resistance, maintaining hyperglycemic levels. The Whole body vibration session may improve the glucose metabolism in diabetic patients by reducing the peripheral blood sugar. Ten healthy elderly women and eight diabetic elderly women were allocated into two groups, and have made an acute whole body session.

ELIGIBILITY:
Inclusion Criteria:

* elderly between 60 to 74 years,
* sedentary according the International Physical Activity Questionnaire (IPAQ- short form)
* For diabetic group, were considered who those medical diagnoses of type II diabetes for at least 02 complete years, who had used only oral hypoglycemic agents of biguanides class (Metformin extended release - XR) in dosage between 500 to 850 mg.
* For healthy elderly group were considered elderly women without self-reported diseases

Exclusion Criteria:

* diabetic volunteers who have ingested the breakfast less than 02 hours or more than 03 hours and those who have taken Metformin less than 02 hours before the intervention.

For all volunteers, the complementary exclusion criteria were:

* the current or past smoking or alcoholic habits;
* the cardiovascular, liver or neuromuscular diseases;
* subjects with prior labyrinthitis or embolic events;
* who have had any surgery in last year;
* volunteers with metallic prosthesis as pacemaker, pins or plates;
* volunteers with advanced osteoporosis;
* which had difficulties during the evaluation or acute protocol.

Ages: 60 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in glucose levels | before and immediately after the 10 minute intervention
  A digital puncture with disposable lancets was collected a peripheral blood drop in the specific strip for the home glucose monitoring AccuChek Active® (Roche Diagnostics GmbH, Mannheim, Germany) according to International Organization for Standardization (ISO) recommendations in 2013 (11).
Changes in lactate levels | before and immediately after the 10 minute intervention
  Another peripheral blood drop was collected from the same digital puncture with disposable lancets and put in the specific strip for to check the seric blood lactate, which was analyzed by a portable lactimeter Accutrend Plus ® (Roche Accutrend Plus, New York, USA).

SECONDARY OUTCOMES:
peripheral oxygen saturation (SpO2) | before and immediately after the 10 minute intervention
  measured with a digital oximeter Onyx (Nonim, model 9500, USA)
heart rate (HR) | before and immediately after the 10 minute intervention
  measured with a digital oximeter Onyx (Nonim, model 9500, USA)
Borg's Rating of Perceived Exertion Scale (RPE) or Modified Borg Scale | before and immediately after the 10 minute intervention
  visual scale that measure the perceived exertion in muscle or dyspnoea, measuring values between 0 at 10

CONTACTS AND LOCATIONS:
Locations (1):
- Maíra F Pessoa, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Undecided